CLINICAL TRIAL: NCT03287843
Title: Effect of Timing of Surgery After Neoadjuvant Chemoradiation on Histopathological Results, Complications, Recurrence and Survivals for Locally Advanced Rectal Cancer
Brief Title: Appropriate Timing of Surgery After Neoadjuvant Chemoradiation for Locally Advanced Rectal Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ege University (Other)
Responsible Party: Principal Investigator, Zekeriya Erhan Akgün, Professor of surgery, Ege University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 17-4.1/13
Record Dates: First submitted 2017-09-13; First posted 2017-09-19 (Actual); Results first posted 2019-08-29 (Actual); Last update posted 2022-03-31 (Actual); Status verified 2022-03

CONDITIONS: Neoplasm, Rectum
Keywords: Locally advanced rectal cancer; Neoadjuvant chemoradiation
MeSH Terms: conditions — Rectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Early surgery group (Experimental): İn this arm patients will go under surgery before eight weeks, after neoadjuvant chemoradiation therapy.
  Interventions: Procedure: Total mesorectal excision before 56 days (4-8 weeks)
- Late surgery group (Experimental): İn this arm patients will go under surgery after eight weeks, after neoadjuvant chemoradiation therapy.
  Interventions: Procedure: Total mesorectal excision after 56 days (8-12 weeks)

INTERVENTIONS:
Procedure: Total mesorectal excision before 56 days (4-8 weeks) — Low anterior resection or abdominoperineal resection
  Arms: Early surgery group
Procedure: Total mesorectal excision after 56 days (8-12 weeks) — Low anterior resection or abdominoperineal resection
  Arms: Late surgery group

SUMMARY:
This study aimed to compare the outcomes of early versus late surgical resection in patients who underwent curative total mesorectal excision after neoadjuvant chemoradiation. Half of the participants will undergo surgery before 8 weeks, while the other half will undergo surgery after 8 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Clinic stage II-III cancer ( T3- T4 tm or/and N(+) disease )
2. Patients with histologically confirmed adenocarcinoma of the rectum
3. Tumor distal border located within 15 cm. from anal verge (as measured by rigid rectoscopy)
4. Standardized total mesorectal excision surgery
5. Tumor must be clinically resectable with curative intent (R0 resection must be most likely)
6. Elective operation
7. The patient must consent to be in the study and the informed consent must be signed

Exclusion Criteria:

1. Clinic stage I and IV cancer disease
2. Patients with malignant disease of the rectum other than adenocarcinoma
3. Recurrent rectal cancer
4. Emergency cases (Mechanical bowel obstruction, perforation)
5. Other previous or concurrent malignancies
6. Any contraindication for radiochemotherapy
7. Previous chemotherapy or radiotherapy to the pelvis
8. Tumor has arisen from chronic inflammatory bowel disease or hereditary polyposis disease
9. American Society of Anesthesiologists Score >3 patients

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 350 (Actual)
Dates: Start 2006-01-01 (Actual); Primary Completion 2017-01-01 (Actual); Study Completion 2022-01-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Z.Erhan Akgun, Proffesor, Principal Investigator — Ege University

REFERENCES:
- [Derived] Akgun E, Caliskan C, Bozbiyik O, Yoldas T, Doganavsargil B, Ozkok S, Kose T, Karabulut B, Elmas N, Ozutemiz O. Effect of interval between neoadjuvant chemoradiotherapy and surgery on disease recurrence and survival in rectal cancer: long-term results of a randomized clinical trial. BJS Open. 2022 Sep 2;6(5):zrac107. doi: 10.1093/bjsopen/zrac107. PMID 36254732
- [Derived] Akgun E, Caliskan C, Bozbiyik O, Yoldas T, Sezak M, Ozkok S, Kose T, Karabulut B, Harman M, Ozutemiz O. Randomized clinical trial of short or long interval between neoadjuvant chemoradiotherapy and surgery for rectal cancer. Br J Surg. 2018 Oct;105(11):1417-1425. doi: 10.1002/bjs.10984. Epub 2018 Aug 29. PMID 30155949

RESULTS

PARTICIPANT FLOW:
Groups:
- Classic Interval Group: İn this arm patients will go under surgery before eight weeks, after neoadjuvant chemoradiation therapy.
  Total mesorectal excision before 56 days (4-8 weeks): Low anterior resection or abdominoperineal resection
- Long Interval Group: İn this arm patients will go under surgery after eight weeks, after neoadjuvant chemoradiation therapy.
  Total mesorectal excision after 56 days (8-12 weeks): Low anterior resection or abdominoperineal resection
Period: Overall Study
Arm/Group | Classic Interval Group | Long Interval Group
Started | 175 | 175
Excluded | 12 (No surgery n=5 R2 resection n=5 Stage IV n=2) | 8 (No surgery n=4 R2 resection n=2 Stage IV n=2)
Lost to Follow up | 3 | 0
Completed | 160 | 167
Not Completed | 15 | 8

BASELINE CHARACTERISTICS:
Population: 350 patients were randomly assigned. After perioperative evaluation of 350 patients who underwent CRT , 15 patients in the CI group (no surgery, 5; R2 resection, 5; stage IV disease, 2; lost to follow-up, 3) and eight in the LI group (no surgery, 4; R2 resection, 2; stage IV disease, 2) were excluded from the study. 327 included in the analysis.
Groups:
- Total: Total of all reporting groups
Arm/Group | Classic Interval Group | Long Interval Group | Total
Number analyzed (Participants) | 160 | 167 | 327
Age, Continuous [Mean (Inter-Quartile Range); unit: years] | 60.4 [22 to 85] | 61.7 [32 to 85] | 61.0 [22 to 85]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 65 | 71 | 136
  Male | 95 | 96 | 191

OUTCOME MEASURES:

1. Primary Outcome: Pathological Complete Response Rate
Description: Complete pathological response, defined as the absence of viable tumor cells, may develop after neoadjuvant treatment for rectal cancer. Prognostic factors affecting pathological complete response will be evaluated.
Time Frame: 2 months
Measure: Count of Participants; unit: Participants
Arm/Group | Classic Interval Group | Long Interval Group
Number analyzed (Participants) | 160 | 167
Participants | 16 | 31

2. Secondary Outcome: Completeness of the Mesorectal Dissection
Description: Examination will be made in a fresh state for completeness of the mesorectal dissection and will be graded according to the criteria of Quirke as follows:
  Low: (Grade 1) Little bulk of the mesorectum with defects down into the muscularis propria and/or very irregular circumferential resection margin.
  Moderate: (Grade 2) Moderate bulk of the mesorectum but there is irregularity in the mesorectal surface. Moderate coning of the specimen toward the distal margin. At no site is the muscularis propria visible with exception of the insertion of the levator muscles. Moderate irregularity of the circumferential resection margin.
  High: (Grade 3) Intact mesorectum with smooth mesorectal surface. No defect deeper than 5 mm. No coning on the specimen. Smooth circumferential resection margins on slicing.
Time Frame: 30 days after surgery
Measure: Count of Participants; unit: Participants
Arm/Group | Classic Interval Group | Long Interval Group
Number analyzed (Participants) | 160 | 167
Participants
  Low | 5 | 8
  Moderate | 11 | 10
  High | 144 | 149

3. Secondary Outcome: Tumour Regression Grade
Description: All pathological examinations were undertaken by two experienced gastrointestinal pathologists. Pathological treatment response to neoadjuvant chemoradiotherapy was evaluated by a five-tiered system described by Mandard.
  Tumor regression grade groups were identified as:
  Grade 1: the absence of residual cancer Grade 2: the presence of residual cancer cells scattered throughout the fibrosis Grade 3: an increase in the number of residual cancer cells but fibrosis still predominant Grade 4: residual cancer outgrowing fibrosis Grade 5, the absence of regressive changes
  Grade 1 considered as complete response. Grade 2-4 considered as partial response and Grade 5 considered as no response.
Time Frame: 30 days after surgery
Measure: Count of Participants; unit: Participants
Arm/Group | Classic Interval Group | Long Interval Group
Number analyzed (Participants) | 160 | 167
Participants
  Mandard Grade 1 | 16 | 31
  Mandard Grade 2 | 37 | 36
  Mandard Grade 3 | 73 | 67
  Mandard Grade 4 | 31 | 29
  Mandard Grade 5 | 3 | 4

4. Secondary Outcome: Surgical Complications
Description: Morbidity will be assessed according to the classification of Clavien-Dindo as follows:
  Grade 1: Any deviation from the normal postoperative course without the need for pharmacological treatment or surgical, endoscopic, and radiological interventions. Allowed therapeutic regimens are: drugs as antiemetics, antipyretics, analgetics, diuretics, electrolytes, and physiotherapy. This grade also includes wound infections opened at the bedside Grade 2: Requiring pharmacological treatment with drugs other than such allowed for grade I complications. Blood transfusions and total parenteral nutrition are also included.
  Grade 3: Requiring surgical, endoscopic or radiological intervention (Grade 3a: Intervention not under general anesthesia, Grade 3b: Intervention under general anesthesia) Grade 4: Life-threatening complication requiring Intensive Care Unit management (Grade 4a: Single organ dysfunction (including dialysis), Grade 4b: Multiorgan dysfunction) Grade 5 Death
Time Frame: 90 days after surgery
Measure: Count of Participants; unit: Participants
Arm/Group | Classic Interval Group | Long Interval Group
Number analyzed (Participants) | 160 | 167
Participants
  Clavien Dindo 1 | 4 | 7
  Clavien Dindo 2 | 15 | 14
  Clavien Dindo 3a | 4 | 3
  Clavien Dindo 3b | 8 | 2
  Clavien Dindo 4a | 4 | 2
  Clavien Dindo 4b | 0 | 1
  Clavien Dindo 5 | 1 | 4
  No complication | 124 | 134

5. Secondary Outcome: Recurrence
Description: Both pelvic recurrence and distant metastasis will be assessed.
Time Frame: 5 years after surgery
Reporting Status: Not Posted

6. Secondary Outcome: Disease-free Survival
Description: Recurrence free survival
Time Frame: 5 years after surgery
Reporting Status: Not Posted

7. Secondary Outcome: Overall Survival
Description: Total survival with or without disease
Time Frame: 5 years after surgery
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | Classic Interval Group | Long Interval Group
All-Cause Mortality (participants affected / at risk) | 1/160 | 4/167
Serious Adverse Events (participants affected / at risk) | 36/160 | 33/167
Other Adverse Events (participants affected / at risk) | 0/160 | 0/167
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Classic Interval Group (N=160) | Long Interval Group (N=167)
Anastomotic leakage (Gastrointestinal disorders) | 4 | 4
Wound infection (Surgical and medical procedures) | 6 | 9
Urinary leakage (Renal and urinary disorders) | 1 | 0
Pelvic abscess (Infections and infestations) | 1 | 2
Postoperative bleeding (Surgical and medical procedures) | 2 | 2
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 | 3
Urinary tract infectio (Renal and urinary disorders) | 3 | 2
Prerenal insufficiency (Renal and urinary disorders) | 5 | 4
Mechanical bowel obstruction (Gastrointestinal disorders) | 5 | 4
Deep vein thrombosis, pulmonary embolism (Vascular disorders) | 2 | 2
Other (Surgical and medical procedures) | 4 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No